CLINICAL TRIAL: NCT00941447
Title: Development of Self-Regulation in Individuals With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Abbott Diabetes Care (Industry)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3R01DK074721 (NIH)
Record Dates: First submitted 2009-07-15; First posted 2009-07-17 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Obesity; Self-Regulation; Self-Efficacy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Self-Control | interventions — Diet; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-Regulation (Experimental): Self Regulation Arm focuses on increasing participants self-monitoring blood glucose (SMBG) AND awareness of self-regulatory approaches to managing diabetes.
  Interventions: Behavioral: Dietary; Behavioral: Physical Activity; Behavioral: Self-Regulatory Approaches
- Self-Monitoring (Experimental): Self-Monitoring Arm focuses on increasing participants self-monitoring blood glucose (SMBG) and providing nutrition education ONLY.
  Interventions: Behavioral: Dietary; Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Dietary — All participants in the investigation will receive a standard 12-week behavioral intervention with seven 30-45 minute phone interventions and education sessions. The intervention includes a reduced caloric prescription (1200-1500 kcal/day),fat gram prescription (30% or less kcals from fat) and carbohydrate gram prescription (150-190 grams).
Behavioral: Physical Activity — There is a physical Activity of 150 minutes/week of moderate-intense physical activity.
Behavioral: Self-Regulatory Approaches — Participants in this arm will receive extensive feedback based on their self-monitoring diary in which the researcher will be reinforced in areas that they are doing well in regarding their blood glucose and also assist in problem solving in areas that need improvement.
  Arms: Self-Regulation

SUMMARY:
The purpose of this investigation is to conduct a 12-week study to compare the effects of a self-regulation intervention (SR), in which participants will self-monitor their blood glucose (BG) and adjust dietary intake and physical activity through the use of current dietary and physical activity guidelines to help regulate their BG, to an education and self-monitoring only intervention (SM), on blood glucose, self-efficacy, and diabetes self-management activities.

DETAILED DESCRIPTION:
As our nation continues to battle overweight and obesity, the prevalence of diabetes will precipitously increase, placing additional financial burden on our country. Therefore, finding ways to manage this chronic disease is essential. While self-monitoring of blood glucose (SMBG) has been shown to be effective in improving glycemic control in individuals with type 1 diabetes, the importance of encouraging individuals with type 2 diabetes to engage in SMBG for better blood glucose (BG) is still unclear. SMBG is believed to be key in the self-management of diabetes, as it can provide feedback on dietary and activity behaviors that are believed to impact on BG. The use of SMBG to adjust other behaviors that impact on BG is a self-regulatory approach to diabetes management. Self-regulation of BG is theorized to impact on self-efficacy in the management of diabetes. Through greater self-efficacy, greater compliance to diabetes self-management behaviors is achieved. Currently, no trial has examined the use of a self-regulation approach using current dietary and physical activity recommendations for individuals with type 2 diabetes who are not on insulin.

Thus, this investigation will involve a 12-week study to examine the effect of an SR intervention to SM intervention. All participants in the investigation will receive a standard 12-week behavioral intervention. The intervention will include a reduced caloric prescription (1200-1500 kcal/day), fat gram prescription (30% or less kcals from fat), carbohydrate gram prescription (150-190 grams/day) and a physical activity goal (slowly building up to 150minutes/week of moderate-intense physical activity at the end of study).

Participants will be assessed at 0 and 13 weeks (pre- and post-intervention) on measures of fasting blood glucose, self-efficacy, and diabetes self-management activities. Additionally, dietary intake, physical activity, quality of life and body weight measurements will be taken at 0 and 13 weeks for comparisons between the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Recruitment from Cherokee Health Systems, Healthy Eating and Activity Laboratory Ineligible Database, UTK faculty and staff, and local endocrinologists' offices.
* Have been diagnosed with Type 2 diabetes for a minimum of 1 year.
* Fasting BG of ≥ 126mg/dl6.
* Between the age of 21 and 65 years. Older adults may have more medical co-morbidities and may require greater medical supervision29.
* Considered overweight or obese by the body mass index (BMI). BMI between 27 and 45 kg/m2 29. The American Diabetes Association 2008 position statement for current nutrition recommendations and interventions for diabetes encourages those individuals within this BMI range to follow the low-calorie, low-fat diet that is prescribed in both conditions in this investigation6.
* Not treated with insulin.
* Are taking medicine that do not typically cause hypoglycemia: Refer to diabetes medication list in Appendices Ai-Aii.
* Willing to increase physical activity to 150mins/week in 3 months.
* Willing to be randomized to either condition.
* Able to report that they can read and understand English.
* Able to report that they can keep a food diary and perform basic mathematics.

Exclusion Criteria:

* Report a heart condition, chest pain during periods of activity or rest or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q). Individuals self-reporting joint problems, prescription medication usage related to heart conditions, or other medical conditions that could limit exercise will be required to obtain written physician consent to participate.
* Report being unable to walk for 2 blocks (1/4 mile) without stopping.
* Report major psychiatric diseases.
* Are compliant with dietary and physical activity recommendations to achieve ideal body weight.
* Taking any weight loss medication.
* Pregnant, expecting to be pregnant and/or lactating.
* Have no working phone.
* Are unwilling to participate in phone calls that are a part of the condition that in which they have been randomized.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Blood Glucose | 12 weeks

SECONDARY OUTCOMES:
Caloric, fat and carbohydrate intake | 12 weeks
Self-efficacy | 12-weeks
Self-management activities | 12 weeks
Physical activities | 12 weeks
Quality of Life | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lusi M Martin, BA, Principal Investigator — University of Tennessee, Knoxville; Hollie A Raynor, Ph.D, Study Chair — University of Tennessee, Knoxville
Locations (1):
- University of Tennessee, Healthy Eating and Activity Laboratory (HEAL), Knoxville, Tennessee, United States